CLINICAL TRIAL: NCT06252896
Title: Investigation Of The Acute Effect Of Device-Assisted Soft Tissue Mobilization Technique on Physical Fitness Parameters In Healthy Individuals
Brief Title: The Acute Effect Of Instrumental-Assisted Soft Tissue Mobilization Technique on Physical Fitness Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Ukbe Sirayder, Sub-Investigator, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/7534Oguz
Record Dates: First submitted 2024-01-12; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Physical Fitness
Keywords: Aerobic Agility; Balance; Capacity; Fatigue; Flexibility; Mobilization
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM Group (Experimental): Individuals were positioned on the stretcher so that the area to be applied was exposed. ADYDM to be applied to ensure comfortable movement of the instrument on the tissue before application baby oil was applied to cover the area. In order to increase the effectiveness of the application suggestions were made to the person to relax. Application ADYDM for each muscle group tool (Figure 3.4) for 5 minutes. The occurrence of allergic reactions on the skin the test was terminated.
  Interventions: Other: INSTRUMENTAL-ASSISTED SOFT TISSUE MOBILIZATION TECHNIQUE
- Control Group (Placebo Comparator): The control group was kept for 30 minutes without ADYDM application and then muscle strength assessment, flexibility assessment, agility assessment, balance assessment and finally aerobic capacity assessment were performed respectively.
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: INSTRUMENTAL-ASSISTED SOFT TISSUE MOBILIZATION TECHNIQUE — After all evaluations were made, IASTM was applied to the individuals in the intervention group for five minutes each, for a total of 20 minutes, on the quadriceps and hamstring muscles of both extremities, respectively.
  Arms: IASTM Group
Other: NO INTERVENTION — The control group waited for 30 minutes after the initial measurements and all measurements were repeated.
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the effect of Instrument Assisted Soft Tissue Mobilization (IASTM) on the acute effects of physical fitness parameters in healthy male individuals. 24 volunteers are included in this study who have been divided into two groups such that one part is an IASTM and the other part is a control group. The physical activity levels of the individuals participating in the study were determined using the short form of the International Physical Activity Assessment Questionnaire (IPAQ). Individuals; their aerobic capacity is the Incremental Shuttle Walk Test (ISWT), muscle strength values are digital dynamometer, muscle flexibility values are sit-reach and quadriceps flexibility test, fatigue values are Fatigue Severity Scale (FSS) and Modified Borg Scale, agility assessment is T-Test, and balance assessment is evaluated with a stabilometer device.

DETAILED DESCRIPTION:
METHOD

Participants

This study was planned as a randomized, parallel-group clinical trial. A total of 24 individuals, 12 in the IASTM group and 12 in the control group were included in the study. We calculated (G*Power Version 3.1.9.4, Franz Faul, Universitat Kiel, Düsseldorf, Germany) a power of 95% with 0.05 significance, a difference to be detected of 6.88 cm, and a standard deviation of 5.22 cm in hamstring flexibility, generating a sample of 12 individuals per group (Figure 1).

Volunteer individuals aged between 18 and 25 years, who could cooperate with the tests and who did not have any diagnosed orthopedic, cardiac, pulmonary, vestibular, and neurological diseases were included in the study. Those who had an allergic reaction during the IASTM application and those who had an acute infection in the last 15 days were excluded. The data were collected from March 2022 to July 2022.

Randomization This study, which was conducted to examine the acute effect of IASTM on physical fitness parameters, was planned as a randomized controlled parallel trial. The sealed envelope method was used for randomization. The procedure was designed by a researcher who was not involved in other aspects of the protocol. All participants were recruited into groups using pre-numbered, sealed, opaque envelopes.

Materials

First, sociodemographic information of all individuals included in the study was obtained, and all questionnaires were conducted.

Hamstring flexibility measurements of the individuals were performed with a sit-and-reach test using a flexibility bench. Quadriceps flexibility was assessed by placing both hips in a neutral position while the subject lay in the prone position.

The Incremental Shuttle Walk Test (ISWT) was performed to assess the exercise capacity of individuals. The test is set to 10 m between two lines for testing. The individual walks a distance of 10 m around the trip and runs as necessary. At the end of the test, the distance traveled by the individual is recorded. Heart rate, blood pressure, oxygen saturation (Cosmed Spiropalm 6MWT, Milan, Italy), respiratory rate, dyspnea, and fatigue level using the modified Borg Scale were evaluated before and after the ISWT.

Muscle strength was determined by measuring quadriceps and hamstring muscle strength using a digital dynamometer (Jtech Commander Muscle Tester, UT, USA). The mean values of the right and left side measurements were obtained. Then, the average of the measurements of the right and left sides were recorded in Newton (N) using each side.

Agility measurements of the cases were made with T-Test. To apply the T-Test, 4 cones were arranged according to the test and the test was performed. Participants had three repetitions and the best time was recorded.

A stabilometer device (HUR Smartbalance 2031, Kokkola, Finland) used in the study is a balance mechanism that can move forward-backward, right-left, and 3D in the transverse plane. The device's reliability has been demonstrated in different studies.

Fatigue levels of individuals were evaluated using the FSS. Our study used the Turkish version of the FSS.

The short form of the International Physical Activity Questionnaire (IPAQ) was used to assess participants' physical activity levels. Severe, moderate-severe, and walking include seven questions that question the time elapsed while doing these, and sitting time is considered a separate question.

Intervention

In this study, the primary outcome measurements were the quadriceps and hamstring flexibility, and the secondary outcome measurements were exercise capacity, muscle strength, agility, balance, and fatigue. The individuals included in the study were divided into two groups: IASTM and control groups. All measurements were performed on individuals in two groups. Then, in the IASTM group, IASTM was applied to the quadriceps and hamstring muscles of both extremities for five minutes each, for a total of 20 minutes. Immediately afterward, the measurements taken before the intervention were repeated. The control group waited for 30 minutes after the initial measurements and all measurements were repeated.

Statistical analyses

Statistical analyses were performed using SPSS Statistics 25.0 (IBM Inc., Armonk, NY, USA). Descriptive statistics were calculated. The normality of the data was checked using the Kolmogorov-Smirnov test. As appropriate, two independent groups of numerical variables were analyzed using Student's t-test or the Mann-Whitney U-test. The chi-square test was used for categorical comparisons. Baseline values were compared using Student's t-test. A two-way analysis of variance was used to evaluate time and group-time interaction. Repeated measures of variance were analyzed in the data in each session. Within-group changes over time were compared using the Wilcoxon signed-rank test. The descriptive level of significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18-25 years,
2. Individuals who volunteered to participate in the study were included.

Exclusion Criteria:

1. Those with diagnosed cardiopulmonary, neurological, orthopedic, psychiatric, skin disease and vestibular diseases,
2. Those who have had an acute infection in the last fifteen days
3. Individuals who showed and/or were at risk of allergic reactions during ADYDM application were not included in the study.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Flexibility | up to six week
  Hamstring flexibility measurements of the individuals were performed with a sit-and-reach test using a flexibility bench. Quadriceps flexibility was assessed by placing both hips in a neutral position while the subject lay in the prone position.

SECONDARY OUTCOMES:
Exercise Capacity | up to six week
  Individuals' exercise capacity will be evaluated using the Incremental Shuttle Walk Test (ISWT), a test that measures maximal aerobic capacity. The test is set to 10 m between two lines for testing. The individual walks a distance of 10 m around the trip and runs as necessary. At the end of the test, the distance traveled by the individual is recorded.
Agility | up to six week
  Agility measurements of the cases were made with T-Test. To apply the T-Test, 4 cones were arranged according to the test and the test was performed. Participants had three repetitions and the best time was recorded.
Balance | up to six week
  A stabilometer device (HUR Smartbalance 2031, Kokkola, Finland) used in the study is a balance mechanism that can move forward-backward, right-left, and 3D in the transverse plane. The device's reliability has been demonstrated in different studies.
Muscle Strength | up to six week
  Muscle strength was determined by measuring quadriceps and hamstring muscle strength using a digital dynamometer (Jtech Commander Muscle Tester, UT, USA). The mean values of the right and left side measurements were obtained. Then, the average of the measurements of the right and left sides were recorded in Newton (N) using each side.
Fatique | up to six week
  Fatigue levels of individuals were evaluated using the Fatigue Severity Scale. Our study used the Turkish version of the FSS.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Kocasinan/Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No